CLINICAL TRIAL: NCT06643468
Title: Evaluation of the Effectiveness of ALB-PRF With Two Types of Bone Grafts With Putty Form in the Treatment of Peri-Implant Bony Defects Around Immediate Dental Implants in the Maxillary Aesthetic Zone.
Brief Title: Effectiveness of ALB-PRF With Two Types of Bone Grafts With Putty Form Around Immediate Dental Implants.
Acronym: ALB-PRFE-PRF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hamzah Abdulatef Mansoor, B.D.S, M.S, Master Degree of Oral Medicine & Periodontology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A02090230M
Record Dates: First submitted 2024-09-22; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dental Implants; Immediate Implant Soft Tissue Healing; Immediate Implant With Bone Graft
Keywords: ALB-PRF; putty form bone graft; e- PRF
MeSH Terms: interventions — Bone Transplantation; beta-tricalcium phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- beta-tricalcium phosphate + calcium sulphate bone graft and collagen membrane (Active Comparator): will include 10 patients, in which participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate as bone graft and collagen as membrane.
  Interventions: Procedure: participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate bone graft and collagen membrane.
- beta-tricalcium phosphate + calcium sulphate bone graft and ALB- PRF membrane (Active Comparator): will include 10 patients, in which participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate as bone graft and ALB- PRF as membrane.
  Interventions: Procedure: participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate bone graft and ALB-PRF membrane.
- nano-crystalline putty hydroxyapatite bone graft and collagen membrane (Active Comparator): will include 10 patients, in which participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and collagen as membrane.
  Interventions: Procedure: participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and collagen membrane.
- nano-crystalline putty hydroxyapatite bone graft and ALB- PRF membrane (Active Comparator): will include 10 patients, in which participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and ALB- PRF as membrane.
  Interventions: Procedure: participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and ALB- PRF as membrane.

INTERVENTIONS:
Procedure: participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and collagen membrane. — 1. Injection of local anesthetic Articaine hydrochloride 4% with Epinephrine (1:100,000).
  2. Atraumatic removal of remaining root or tooth then implant will be placed according to the standard protocol.
  3. Sulcular incision with be made 15c blade .
  4. Implant placement with copious irrigation.
  5. Membranes placement: collagen followed by insertion of nano-crystalline putty hydroxyapatite.
  6. Customized healing abutment application.
  7. Suturing of wound edges with 0.5 suture around the customized healing abutment.
  Arms: nano-crystalline putty hydroxyapatite bone graft and collagen membrane
Procedure: participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and ALB- PRF as membrane. — 1. Injection of local anesthetic Articaine hydrochloride 4% with Epinephrine (1:100,000).
  2. Atraumatic removal of remaining root or tooth then implant will be placed according to the standard protocol.
  3. Sulcular incision with be made 15c blade without vertical releasing incision.
  4. Implant placement with copious irrigation.
  5. Membranes placement: ALB-PRF followed by insertion of nano-crystalline putty hydroxyapatite..
  6. Customized healing abutment application.
  7. Suturing of wound edges with 0.5 suture around the customized healing abutment.
  Arms: nano-crystalline putty hydroxyapatite bone graft and ALB- PRF membrane
Procedure: participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate bone graft and collagen membrane. — 1. Injection of local anesthetic Articaine hydrochloride 4% with Epinephrine (1:100,000).
  2. Atraumatic removal of remaining root or tooth then implant will be placed according to the standard protocol.
  3. Sulcular incision with be made 15c blade .
  4. Implant placement with copious irrigation.
  5. Membranes placement: collagen followed by insertion of eta-tricalcium phosphate + calcium sulphate bone graft.
  6. Customized healing abutment application.
  7. Suturing of wound edges with 0.5 suture around the customized healing abutment.
  Arms: beta-tricalcium phosphate + calcium sulphate bone graft and collagen membrane
Procedure: participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate bone graft and ALB-PRF membrane. — 1. Injection of local anesthetic Articaine hydrochloride 4% with Epinephrine (1:100,000).
  2. Atraumatic removal of remaining root or tooth then implant will be placed according to the standard protocol.
  3. Sulcular incision with be made 15c blade .
  4. Implant placement with copious irrigation.
  5. Membranes placement: ALB-PRF followed by insertion of eta-tricalcium phosphate + calcium sulphate bone graft.
  6. Customized healing abutment application.
  7. Suturing of wound edges with 0.5 suture around the customized healing
  Arms: beta-tricalcium phosphate + calcium sulphate bone graft and ALB- PRF membrane

SUMMARY:
The goals of this clinical trial study is to evaluate the additive effect, of using ALB-PRF membrane combined with two different types of bone grafts with putty form in treatment of peri-implant bony defects around immediate dental implant within the maxillary esthetic zone.

Researchers will compare the ALB- PRF membrane extracted from patient blood with synthetic collagen membrane in addition to the putty form bone graft The main questions it aims to answer are:

Is the ALB-PRF is considered suitable alternative to synthetic collagen membrane in GBR techniques? also, growth factors releasing form ALB-PRF can continue over 21 days.

Participants will:

receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and collagen as membrane. Also, in other hand participant will receive immediate implant with beta-tricalcium phosphate + calcium sulphate as bone graft and collagen as membrane. and compered with participants receive the same bone and implant technique except for ALB-PRF membrane instead of collagen.

DETAILED DESCRIPTION:
I) Patient selection Participants will be selected from the outpatient clinic in the Oral Medicine and Periodontology Department, Faculty of Dentistry, Mansoura University. All patients will be informed regarding the study nature of the surgical procedures, time of treatment, benefits, the suspected risk or complications and follow-up schedule visits and requested to sign a written consent. This study will be performed after getting approval by the ethics committee of the Faculty of Dentistry at Mansoura University.(A02090230M)

Inclusion criteria:

* Patient between 20-40 years old.
* Unrestorable maxillary tooth/ teeth in the aesthetic zone.
* Adequate keratinized soft tissue.
* Favorable pattern of occlusion.
* Good oral hygiene.
* Patient ability to comply with the required recall visits.
* Patients with type II socket.

Exclusion Criteria:

* Local or systemic diseases that contraindicate implant placement or surgery.
* Smokers
* Patients with parafunctional habits.

Study design:

Selected participants will receive forty implants that will be placed immediately after extraction of unrestorable maxillary tooth/ teeth in the aesthetic zone. According to the type of the used bone graft and membrane, the participants will be randomly divided into 4 equal groups:

Group I: will include 10 patients, in which participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and collagen as membrane. Group II: will include 10 patients, in which participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate as bone graft and collagen as membrane.

Group III: will include 10 patients, in which participants will receive immediate implant with nano-crystalline putty hydroxyapatite as bone graft and ALB- PRF as membrane. Group IV: will include 10 patients, in which participants will receive immediate implant with beta-tricalcium phosphate + calcium sulphate as bone graft and ALB- PRF as membrane.

Procedures:

Pre-surgical phase:

* Pre-operative CBCT will be used to evaluate the mesiodistal width (inter-radicular distance), residual bone beyond the apex, socket width and root angulation.
* Study cast analysis to evaluate teeth inclinations, inter-arch space and occlusion. - Diagnostic waxing up of missing tooth.
* Premedication: Patients will be premedicated by Amoxicillin 2 gm one hour before surgery as a prophylactic antibiotic, in addition patient will instructed to rinse with a 0.2% chlorhexidine mouth wash for 1 minute immediately prior to surgery.

Surgical phase:

1. Injection of local anesthetic Articaine hydrochloride 4% with Epinephrine (1:100,000).
2. Atraumatic removal of remaining root or tooth then implant will be placed according to the standard protocol.
3. Sulcular incision with be made 15c blade Minimally vertical releasing incision.
4. Implant placement with copious irrigation.
5. Membranes placement: either ALB-PRF or collagen followed by insertion of putty form of bone graft materials according to the study design.
6. Customized healing abutment application.
7. Suturing of wound edges with 0.5 suture around the customized healing abutment.

Post-surgical instruction:

* Patients will be instructed to use 0.2% chlorhexidine gluconate mouth wash for 1 minute twice a day for 2 weeks.
* Patients will be maintained on amoxicillin 1gm twice a day for six days postoperatively.
* Ibuprofen 400 mg will be prescribed to be taken 2 to 4 times a day during meals as analgesic.

Loading on implant will be done four months after the implant insertion.

Evaluation:

I) Clinical Evaluation: all the following clinical parameters will be reassessed at 0,6,12 months.

1. Esthetics:

   Will be evaluated according to pink esthetic score (PES).
2. Peri-implant pocket depth:

   The distance between the base of the pocket and the gingival margin will be measured using a graduated plastic probe.
3. Plaque index (PI) :

   Plaque index will be taken as an indicator for the patient oral hygiene.
4. Implant stability evaluation:

   Using Resonance Frequency Analysis device (Osstell), implant stability will be assessed in both groups at baseline, 6 months , and 12 months postoperative
5. Modified bleeding index. Modified bleeding index will be taken as an indicator gingival inflammation.

II) Radiographic Evaluation:

Using cone beam CT (CBCT) scan, the changes in the marginal bone level and the thickness of buccal plate will be measured at baseline, 6 months and 12 months postoperative.

III) Laboratory analysis :

Samples will be collected using sterile paper strip at day of surgery, one, two, four, and eight weeks postoperatively for analysis of the growth factors concentration according to manufacture instruction using multiplex immunoassay.

Statistical analysis:

The data will be collected and statistical analysis will be done

ELIGIBILITY:
Inclusion Criteria:

* - Patient between 20-40 years old.
* Unrestorable maxillary tooth/ teeth in the aesthetic zone.
* Adequate keratinized soft tissue.
* Favorable pattern of occlusion.
* Good oral hygiene.
* Patient ability to comply with the required recall visits.
* Patients with type II socket.

Exclusion Criteria:

* Local or systemic diseases that contraindicate implant placement or surgery.
* Smokers
* Patients with parafunctional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
soft tissue healing. in relation to different membrane and putty form bone | clinical parameters will be reassessed at plate will be measured at baseline, 6 months and 12 months postoperative.
  Evaluate if the ALB-PRF membrane in combination with the two tested putty form bone graft materials play a role in acceleration of soft tissues healing.
  assessment of soft tissue healing which evaluated according to pink esthetic score (PES).
  The pink esthetic score evaluates the esthetic outcome of soft tissue around implant-supported single crowns in the anterior zone by awarding seven points for the mesial and distal papilla, soft-tissue level, soft-tissue contour, soft-tissue color, soft-tissue texture, and alveolar process deficiency. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value, the maximum achievable PES was 14
Hard tissue healing . | baseline, 6 months and 12 months postoperative
  Hard tissue healing evaluation; Using cone beam CT (CBCT) scan, the changes in the marginal bone level and the thickness of buccal plate will be measured at baseline, 6 months and 12 months postoperative.
  CBCT will be evaluated and assessed by subtraction methods to notice the gained and loosed bone in millimeters.

SECONDARY OUTCOMES:
Peri-implant pocket depth | baseline, 6 months and 12 months postoperative.
  The distance between the base of the pocket and the gingival margin will be measured using a graduated plastic probe.
Implant stability evaluation | baseline, 6 months , and 12 months postoperative
  Using Resonance Frequency Analysis device (Osstell®), implant stability will be assessed in both groups
Modified bleeding index | baseline, 6 months , and 12 months postoperative
  Modified bleeding index will be taken as an indicator gingival inflammation.
growth factors concentration | one, two, four, and eight weeks postoperatively
  Samples will be collected using sterile paper strip at day of surgery, one, two, four, and eight weeks postoperatively for analysis of the growth factors concentration according to manufacture instruction using multiplex immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Mansoura university ,, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
after Completing the study ; the data will be available when requested